CLINICAL TRIAL: NCT03010969
Title: Perioperative Endothelial Dysfunction in Patients Undergoing Major Acute Abdominal Surgery. The POETRY Abdominal Study
Brief Title: Perioperative Endothelial Dysfunction in Patients Undergoing Major Acute Abdominal Surgery
Acronym: POETRYabd
Status: Completed | Type: Observational
Sponsor: Zealand University Hospital (Other)
Responsible Party: Principal Investigator, Sarah Victoria Ekeløf Busch, MD, Zealand University Hospital
Other Study IDs: POETRY abdominal
Record Dates: First submitted 2016-12-16; First posted 2017-01-05 (Estimated); Last update posted 2021-02-17 (Actual); Status verified 2021-02

CONDITIONS: Cardiovascular Complication; Complication, Postoperative
Keywords: Endothelial dysfunction; Surgery; Pulmonary function; Blood glucose level; Patient-related outcomes
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The blood will be collected from a larger vein (e.g. the cubital vein). Cardiac troponin I Tetrahydrobiopterin: Blood is sampled into 4mL EDTA tubes. Immediately after withdrawal, a minimum of 1mL blood is mixed with 25μL DTE. The mixture is centrifuged at 2000g for 5 minutes. Plasma is frozen and stored at -80°C.
  Arginine and ADMA: Blood is sampled into 4mL EDTA tubes. Blood samples will be centrifuged at 3000g for 10 minutes, plasma frozen and stored at -80°C until analyzed with high performance liquid chromatography.
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Acute abdominal surgery — Acute abdominal surgery within 72 hours of admission to the department of surgery

SUMMARY:
The aim of the clinical study is:

1. to examine the association between postoperative endothelial function, indirectly measured by reactive hyperemia index, and major adverse cardiovascular events including myocardial injury and cardiac death within 30, 90 and 365 days of acute abdominal surgery.
2. to examine the association between postoperative endothelial function, indirectly measured by reactive hyperemia index, and non-cardiovascular complications including non-cardiac death within 30, 90 and 365 days of acute abdominal surgery.
3. to examine the importance of the postoperative blood glucose level and the pulmonary function for postoperative complications and death within 30, 90 and 365 days of acute abdominal surgery.
4. to examine the association between postoperative endothelial function, pulmonary function and blood glucose level
5. the qualitative part of the study will examine the postoperative subjective symptoms including acute and chronic pain, quality of recovery and functional status, depressive thoughts and post-traumatic stress disorder.

ELIGIBILITY:
Inclusion criteria

* ≥ 18 years old
* Surgery within 72 hours of an acute admission to the Department of Surgery or an acute reoperation.
* Major gastrointestinal surgery on the gastrointestinal tract. This will include
* Open, laparoscopic, or laparoscopically-assisted procedures
* Procedures involving the stomach, small or large bowel, or rectum for conditions such as perforation, ischaemia, abdominal abscess, bleeding or obstruction
* Washout/evacuation of intra-peritoneal abscess (unless due to appendicitis or cholecystitis - excluded, see below)
* Washout/evacuation of intra-peritoneal hematoma
* Bowel resection/repair due to incarcerated umbilical, inguinal and femoral hernias (but not hernia repair without bowel resection/repair)
* Bowel resection/repair due to obstructing/incarcerated incisional hernias provided the presentation and findings were acute
* Laparotomy/laparoscopy with inoperable pathology (e.g. peritoneal/hepatic metastases)
* Laparoscopic/Open Adhesiolysis
* Return to theatre for repair of fascial dehiscence
* Any reoperation/return to theatre meeting the criteria above is included

If multiple procedures (primary surgery or reoperation) are performed on different anatomical sites within the abdominal/pelvic cavity, the patient would be included if the major procedure is general surgical.

Exclusion criteria

* Not capable of giving informed consent after oral and written information
* Previously included in the trial
* If transferred directly from the operation room or recovery ward to the intensive care unit
* Elective laparoscopy
* Diagnostic laparotomy/laparoscopy where no subsequent procedure is performed (NB, if no procedure is performed because of inoperable pathology, then include)
* Appendectomy +/- drainage of localized collection unless the procedure is incidental to a non-elective procedure on the GI tract
* Cholecystectomy +/- drainage of localized collection unless the procedure is incidental to a non-elective procedure on the GI tract (All surgery involving the appendix or gallbladder, including any surgery relating to complications such as abscess or bile leak is excluded)
* Non-elective hernia repair without bowel resection.
* Minor abdominal wound dehiscence unless this causes bowel complications requiring resection
* Ruptured ectopic pregnancy, or pelvic abscesses due to pelvic inflammatory disease
* Laparotomy/laparoscopy for pathology caused by blunt or penetrating trauma
* Laparotomy/laparoscopy for esophageal pathology Laparotomy/laparoscopy for pathology of the spleen, renal tract, kidneys, liver, gall bladder and biliary tree, pancreas or urinary tract

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing major acute gastrointestinal surgery
Sampling Method: Probability Sample
Enrollment: 224 (Actual)
Dates: Start 2016-10; Primary Completion 2018-11 (Actual); Study Completion 2019-11 (Actual)

PRIMARY OUTCOMES:
The change in reactive hyperemia index assessed by EndoPat | The change from 4-24 hours to between day 3 and 5 after surgery
Major adverse cardiovascular events | Within 365 days of surgery
  * Cardiovascular death
  * Myocardial injury within postoperative day 3 (definition: peak plasma cardiac troponin-I ≥ 45ng/L (99th percentile URL, 10% CV at 40ng/L))
  * Acute coronary syndrome (unstable angina pectoris, NSTEMI, STEMI)
  * Congestive heart failure
  * Stroke
  * Nonfatal cardiac arrest
  * New clinically important cardiac arrhythmia
  * Coronary revascularization procedure (PCI or CABG)
  * Sudden unexpected death
Postoperative non-cardiovascular complications | Within 365 days of surgery
  Non-cardiovascular death, sepsis, pneumonia, respiratory failure, surgical complications (min. Clavien-Dindo stage 3), Any non-cardiovascular life-threatening complication (Clavien-Dindo stage 4).

SECONDARY OUTCOMES:
Nitric oxide biomarkers | 4-24 hours after surgery and between postoperative day 3-5
Reactive hyperemia index assessed by EndoPat | 4-24 hours after surgery
Reactive hyperemia index assessed by EndoPat | between day 3 and 5 after surgery
Blood Glucose level | Postoperative day 1 - 7 (or until discharge)
Pulmonary function | Postoperative day 1 - 7 (or until discharge)
Readmission | Readmissions within 1 year of discharge
Lengths of stay | Lengths of stay from the operation day to discharge, on average 14 days.
Lengths of stay in the intensive care unit | Lengths of stay from the operation day to discharge from hospital, on average 14 days.

OTHER OUTCOMES:
Postoperative quality of recovery (QoR15) | postoperative day 1, 3, 5, 7, 14, 30, 90 and 365
  QoR15 score
Numerical rating scale (NRS) pain score | postoperative day 1, 3, 5, 7, 14, 30, 90 and 365
  NRS pain score in rest and at activity
Post-Traumatic Stress Disorder | postoperative day 14, 30, 90 and 365
  Post-Traumatic Stress Disorder questionnaire
Depressive thoughts | postoperative day 14, 30, 90 and 365
  Hospital anxiety and depression scale
Postoperative pain | postoperative day 14, 30, 90 and 365
  Questionnaire Self-reported Leeds Assessment of Neuropatic Symptoms and Signs pain scale (S-LANSS)
Functional status | postoperative day 14, 30, 90 and 365
  Activity Assessment Scale

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Ekeloef, MD, Principal Investigator — Department of Surgery, Zealand University Hospital; Jakob Burcharth, MD, Phd., Principal Investigator — Department of Surgery, Zealand University Hospital
Locations (1):
- Department of Surgery, Zealand University Hospital, Koge, Køge, Denmark

IPD SHARING:
Plan to Share IPD: No
We do not plan to share IPD

REFERENCES:
- [Derived] Ekeloef S, Oreskov JO, Falkenberg A, Burcharth J, Schou-Pedersen AMV, Lykkesfeldt J, Gogenur I. Endothelial dysfunction and myocardial injury after major emergency abdominal surgery: a prospective cohort study. BMC Anesthesiol. 2020 Mar 16;20(1):67. doi: 10.1186/s12871-020-00977-0. PMID 32178626